CLINICAL TRIAL: NCT06589206
Title: Three-Dimensional Assessment of Dentoskeletal Changes Associated With a Modified Twin Block Appliance for Treatment of Skeletal Class II Growing Patients With Mandibular Deficiency: A Randomized Clinical Trial
Brief Title: Three-Dimensional Assessment of Dentoskeletal Changes Associated With a Modified Twin Block Appliance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aml Saeed Mohamed Abdel qader, Lecturer Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3444
Record Dates: First submitted 2024-08-24; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Growth Modification
Keywords: twin block; esthetic twin block; clear twin block; Deficient mandible; Skeletal Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional twin block (Active Comparator): Growing patients with class II skeletal discrepancy due to mandibular deficiency will be treated with the conventional design of twin block previously introduced by Clark.
  Interventions: Other: modified design of twin block
- Vacuum formed twin block appliance with sagittal blocks (Experimental): Growing patients with class II skeletal discrepancy due to mandibular deficiency will be treated with a modified design of twin block formed of vacuum sheets with sagittal blocks.
  Interventions: Other: modified design of twin block

INTERVENTIONS:
Other: modified design of twin block — Vacuum formed twin block appliance with sagittal blocks

SUMMARY:
The aim of the current study is to evaluate the skeletal, dental, soft tissue, TMJ, and upper airway size changes associated with a new design of twin block compared to the conventional twin block appliance. Additionally, patients' satisfaction with the two designs will be assessed.

DETAILED DESCRIPTION:
Twin block appliance is the gold standard for the treatment of skeletal class II patients with deficient mandible. Yet, it has some drawbacks as proclination of the mandibular incisors, development of posterior open bite and the unesthetic appearance. Many modifications in twin block A new design were made to overcome the previous problems, as adding incisor capping, Clasps, sagittal blocks, and esthetic twin block appliances. In the current trial A new design of esthetic twin block appliance with sagittal blocks is investigated and the post treatment skeletal, dental, and soft tissue, TMJ, and upper airway size will be assessed and compared to the changes associated with the conventional design of twin block. Moreover, patient satisfaction with the appliance will be assessed with both appliances.

ELIGIBILITY:
Inclusion Criteria:

* skeletal class II deficient mandible
* Class II molar and canine relation
* male growing patients CVM 2,3 age range 10-14
* normal vertical growth pattern
* ANB > 4
* mild to moderate crowding

Exclusion Criteria:

* Previous orthodontic treatment.
* Craniofacial syndrome.
* Periodontal disease.
* Extracted first permanent molars.

Ages: 10 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
skeletal changes | 9 months
  changes in SNA, SNB, and ANB angles will be measured before and after treatment
Dental changes | 9 months
  changes in maxillary and mandibular incisors position and inclination will be assessed before and after treatment

SECONDARY OUTCOMES:
soft tissue changes | 9 months
  changes in soft tissue A, B, Pog points will be assessed before and after treatment
JMJ changes | 9 months
  changes in the TMJ morphologic structure will be assessed before and after treatment
Upper airway size | 9 months
  changes in the Upper airway size will be assessed before and after treatment
patient satisfaction | after one and nine months
  patients acceptance of the appliance will be assessed by a questionnaire administered in one to one interview.